CLINICAL TRIAL: NCT00200746
Title: Arginine Treatment for Alcoholic Hepatitis
Brief Title: Treatment of Alcohol-Related Hepatitis With Arginine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Responsible Party: John Tayek, M.D., La BioMedical
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21AT002394-01A1 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Alcoholic Hepatitis
Keywords: Hepatitis; Liver Diseases; Alcoholism; Arginine
MeSH Terms: conditions — Hepatitis, Alcoholic; Hepatitis; Liver Diseases; Alcoholism | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): Moderate Arginine
  Interventions: Drug: Arginine
- 3 (Sham Comparator): Polycose control arm
  Interventions: Drug: Arginine
- 1 (Experimental): High Arginine
  Interventions: Drug: Arginine

INTERVENTIONS:
Drug: Arginine — Amino Acid Arginine

SUMMARY:
The purpose of this study is to test the effectiveness of the amino acid arginine in reducing liver injury in individuals with alcohol-related hepatitis.

DETAILED DESCRIPTION:
Arginine is a naturally occurring amino acid that is also available in pill form. Arginine pills have been shown to aid in liver detoxification and fat breakdown in the liver. Numerous studies have examined the effects of arginine on the liver. However, few have determined the optimal concentration of arginine that would best prevent injury to the liver This study will provide participants with three concentration levels of arginine to determine which is most effective in reducing liver injury in alcoholic hepatitis patients.

This study will last 31 days. Participants will be admitted to the General Clinical Research Center for 27 days. Participants will be randomly assigned to one of four groups. Participants in Groups 1, 2, and 3 will have 1%, 2%, or 6% arginine added to their diet in the form of gel capsules. Participants in Group 4 will receive placebo capsules. Participants will be given 24 capsules of different dietary supplements, including the arginine supplements, every day during their hospital stay.

Participants who are not able to ingest at least 18 capsules per day over 3 days or who are not able to eat the majority of their solid or liquid diet while hospitalized will have a naso-gastric soft feeding tube inserted for food and supplements to be administered. A liver biopsy will be performed on Days 3 and 26. The biopsies will involve insertion of a catheter in a neck vein and a small sample of liver tissue will be removed. On Days 2 and 25, participants will undergo blood and urine collection. Participants will also be infused with nonradioactive leucine to determine the levels of albumin, a protein that is reduced in diseased livers. If participants develop fluid in the abdomen (a condition known as ascites), a small sample of fluid will be extracted from the abdomen twice a day on Days 2, 17, and 25. On Day 31, participants will return to the research center for additional blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcoholic hepatitis
* Maddrey's DF score less than 33

Exclusion Criteria:

* Hepatitis C or B virus infected
* HIV infected
* History of cancer
* Hepatic encephalopathy (a condition in which liver failure affects the central nervous system)
* Kidney failure
* A Do Not Resuscitate order (a patient-directed order not to resuscitate in the event that resuscitation is necessary to prevent death)
* Maddrey's DF score of 33 or greater after vitamin K administration during the study
* Alcohol withdrawal at study entry
* Active pneumonia at study entry
* Allergy to iodine
* Enrollment in any other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percent reduction in liver endotoxin production | After nutritional intervention
change in Maddrey's discriminant function (DF) score | After nutritional intervention

CONTACTS AND LOCATIONS:
Overall Officials: John A. Tayek, MD, Principal Investigator — Los Angeles Biomedical Research Institute at Harbor - University of Los Angeles Medical Center
Locations (1):
- Harbor - University of California Los Angeles Medical Center, Torrance, California, United States